CLINICAL TRIAL: NCT02897479
Title: A Phase II, Open-label Study to Evaluate the Efficacy and Safety of HMPL-504 in Locally Advanced/Metastatic MET-Mutation-Positive Pulmonary Sarcomatoid Carcinomas and Other Non-small Cell Lung Cancer
Brief Title: A Phase II Study of HMPL-504 in Lung Sarcomatoid Carcinoma and Other Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-504-00CH1
Record Dates: First submitted 2016-08-29; First posted 2016-09-13 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-08

CONDITIONS: Lung Sarcomatoid Carcinoma
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Savolitinib (Experimental): Pulmonary Sarcomatoid Carcinomas
  Interventions: Drug: Savolitinib

INTERVENTIONS:
Drug: Savolitinib — Enrolled patients will be treated with Savolitinib 600mg or 400mg once per day(QD), till disease progression, death or unacceptable toxicity, whichever comes first. A cycle of study treatment will be defined as 21 days of continuous dosing.
  Other Names: hmpl-504

SUMMARY:
This is a Phase II, open-label, multicenter study of Savolitinib administered orally once per day(QD) to locally advanced/metastatic PSC patients and other NSCLC patients with MET Exon 14 mutation. The targeted population is the patients with MET Exon 14 mutation who have failed prior systemic therapy (ies), or are unwilling or can not tolerate to receive chemotherapy. Pathological diagnosis will be confirmed retrospectively by the central pathological laboratory.

DETAILED DESCRIPTION:
Savolitinib will be administrated 600mg or 400mg once per day (QD). The treatment will be discontinued for the patients who experience disease progression, death or experience unacceptable toxicity, whichever occurs first. A cycle of study treatment will be defined as 21 days of continuous dosing.

ELIGIBILITY:
Inclusion Criteria:

* 1.Fully understood the study and voluntarily signed Informed Consent Form
* 2.Age > 18 years
* 3.Histologically or cytologically documented locally advanced or Metastatic pulmonary sarcomatoid carcinoma (PSC) patients and other Non-small cell lung cancer（NSCLC） with MET Exon 14 mutation who have failed piror systemic therapy(ies), or are unwilling or unable to receive chemotherapy
* 4.Patient should have measurable disease per RECIST1.1
* 5.ECOG performance status of 0, or 1
* 6.Expected survival > 12 weeks

Exclusion Criteria:

* 1.Co-existing malignancy or malignancies diagnosed within the last 3 years other than lung cancer with the exception of adequately treated skin basal cell carcinoma or cervical cancer in situ.
* 2.Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy or radiotherapy within 3weeks prior to initiation of study treatment, or received TKI (for ex. EGFR-TKI) treatment within 2 week prior to initiation of study treatment
* 3.Palliative radiation to bone metastases within 2 weeks prior to the initiation of study treatment
* 4.Herbal therapy within 1 week prior to the initiation of study treatment
* 5. has EGFR, ALK or ROS 1 positive mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess objective response rate (ORR) | 1year
  ORR is defined as the proportion of patients with complete response or partial response. The confirmation of response for patients who has PR or CR at first time should be performed by at least 4 weeks and in this study, it could be performed by the scheduled tumor assessment 6 weeks later

SECONDARY OUTCOMES:
Progression free survival(PFS) | 1year
  PFS is defined as the Progression free surviva of patients with complete response or partial response or stable disease. In the case of SD, measurements must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks.
Safety Assessment Parameter | 1year
  The safety will be assessed using the following safety outcome measures: incidence of adverse events, physical examinations,vital signs and laboratory tests (including hematology, clinical chemistry, urine tests and other indicators)12-ECG parameters and echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Shun LU, doctor, Principal Investigator — Shanghai Chest Hospital
Locations (2):
- China (2):
  - Beijing Cancer Hopspital, Beijing, Beijing Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu Y, Ren Y, Fang J, Cao L, Liang Z, Guo Q, Han S, Ji Z, Wang Y, Sun Y, Chen Y, Li X, Xu H, Zhou J, Jiang L, Cheng Y, Han Z, Shi J, Chen G, Ma R, Fan Y, Sun S, Jiao L, Jia X, Wang L, Lu P, Xu Q, Luo X, Su W, Lu S. Circulating tumour DNA biomarkers in savolitinib-treated patients with non-small cell lung cancer harbouring MET exon 14 skipping alterations: a post hoc analysis of a pivotal phase 2 study. Ther Adv Med Oncol. 2022 Oct 31;14:17588359221133546. doi: 10.1177/17588359221133546. eCollection 2022. PMID 36339926
- [Derived] Paik PK, Pfeiffer BM, Vioix H, Garcia A, Postma MJ. Matching-Adjusted Indirect Comparison (MAIC) of Tepotinib with Other MET Inhibitors for the Treatment of Advanced NSCLC with MET Exon 14 Skipping Mutations. Adv Ther. 2022 Jul;39(7):3159-3179. doi: 10.1007/s12325-022-02163-9. Epub 2022 May 11. PMID 35543963
- [Derived] Lu S, Fang J, Li X, Cao L, Zhou J, Guo Q, Liang Z, Cheng Y, Jiang L, Yang N, Han Z, Shi J, Chen Y, Xu H, Zhang H, Chen G, Ma R, Sun S, Fan Y, Li J, Luo X, Wang L, Ren Y, Su W. Once-daily savolitinib in Chinese patients with pulmonary sarcomatoid carcinomas and other non-small-cell lung cancers harbouring MET exon 14 skipping alterations: a multicentre, single-arm, open-label, phase 2 study. Lancet Respir Med. 2021 Oct;9(10):1154-1164. doi: 10.1016/S2213-2600(21)00084-9. Epub 2021 Jun 21. PMID 34166627